CLINICAL TRIAL: NCT02095613
Title: A Randomized Trial of Ready-to-use-supplementary Food Compared to Corn-soy-blend+ as Food Rations for HIV-infected Adults on Antiretroviral Therapy in Rural Haiti
Brief Title: Tailored Nutrition and Food Security Interventions in Comprehensive HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Partners in Health (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Louise Ivers, MD, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008P002017/BWH; R01HD057627 (NIH)
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: HIV; Food Insecurity; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corn-soy-blend plus (Active Comparator): food A type of ground meal called corn-soy-blend plus
  Interventions: Other: traditional food
- Ready-to-use-supplementary food (Active Comparator): food A nutrient dense food comprised of peanuts, oil, multivitamins.
  Interventions: Other: food that is nutrient dense

INTERVENTIONS:
Other: traditional food
  Arms: Corn-soy-blend plus
Other: food that is nutrient dense
  Arms: Ready-to-use-supplementary food

SUMMARY:
The study hypothesizes that one form of food supplement to HIV-infected individuals in Haiti (ready-to-use-supplementary food) will result in improved HIV, nutrition and quality of life outcomes when compared to a second type of food supplement (corn-soy-blend) over the course of 12 months of food supplementation.

ELIGIBILITY:
Inclusion Criteria:

* documented to have HIV infection by standard laboratory procedures
* live in the geographic catchment area of PIH services where study is taking place
* 18 years of age or older
* started antiretroviral therapy for HIV in the 24 months prior to study enrollment

Exclusion Criteria:

* if another household member is also eligible for food assistance
* if subject is pregnant at the time of enrollment
* if unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index over time | 6-month, 12-month

SECONDARY OUTCOMES:
Change in Quality of Life over time | 6-month, 12-month

OTHER OUTCOMES:
Change in CD4 cell count over time | 6-month, 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Louise Ivers, MB, BCh, BAO, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Zanmi Lasante, Marc, Haiti